CLINICAL TRIAL: NCT05310747
Title: Can Exposure to Inclusive Virtual Art Decrease Pain and Social Disconnection Among Individuals Living With Chronic Pain?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 1811205
Record Dates: First submitted 2021-12-16; First posted 2022-04-05 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain; Social Disconnection
Keywords: Pain; Social Disconnection; Museum; Virtual museum
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Intervention Model Description: Eligible individuals will be randomized to one of 4 groups:
  1. Artwork present + Social connection prime high
  2. Artwork present + Social connection prime low
  3. Artwork absent + Social connection prime high
  4. Artwork absent + Social connection prime low
  5. Hanging control group - no exposure to any independent variables (i.e. artwork: present or absent; social connection prime: high or low)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Artwork present + social connection high (Experimental): Individuals participate in an exercise to prime a feeling of high social connection and then explore a virtual museum exhibit with artwork for 10 minutes
  Interventions: Behavioral: Artwork present; Behavioral: Social connection high
- Artwork present + social connection low (Experimental): Individuals participate in an exercise to prime a feeling of low social connection and then explore a virtual museum exhibit with artwork for 10 minutes
  Interventions: Behavioral: Artwork present; Behavioral: Social connection low
- Artwork absent + social connection high (Experimental): Individuals participate in an exercise to prime a feeling of high social connection and then explore a virtual museum exhibit with no artwork for 10 minutes
  Interventions: Behavioral: Artwork absent; Behavioral: Social connection high
- Artwork absent + social connection low (Active Comparator): Individuals participate in an exercise to prime a feeling of low social connection and then explore a virtual museum exhibit with no artwork for 10 minutes
  Interventions: Behavioral: Artwork absent; Behavioral: Social connection low
- Hanging control group (No Intervention): Individuals will receive no exposure to any independent variables (i.e. artwork: present or absent; social connection prime: high or low) for 10 minutes before completing their final survey.

INTERVENTIONS:
Behavioral: Artwork present — A virtual museum exhibit with a curated selection of artworks
  Arms: Artwork present + social connection high; Artwork present + social connection low
Behavioral: Artwork absent — The same virtual museum exhibit space as the 'Artwork present' condition but with all of the artworks removed from the walls
  Arms: Artwork absent + social connection high; Artwork absent + social connection low
Behavioral: Social connection high — Participants will identify a person from their life that makes them feel socially connected and then write (1) about that person and (2) an experience they had with that person that made them feel socially connected.
  Arms: Artwork absent + social connection high; Artwork present + social connection high
Behavioral: Social connection low — Participants will identify a person from their life that makes them feel socially disconnected and then write (1) about that person and (2) an experience they had with that person that made them feel socially disconnected.
  Arms: Artwork absent + social connection low; Artwork present + social connection low

SUMMARY:
The proposed study is an experimental intervention to test for the effects of exposure to art by means of a virtual museum visit. It examines the fundamental question of whether exposure to virtual art can alleviate pain. Google Arts & Culture has digitized the collections of over 2,000 museums, art galleries, and other cultural institutions. The platform is free and allows 'visitors' to explore art from around the world. For this study, the PIs have chosen artwork from this collection and created a virtual museum gallery such that research participants will visit the museum with or without art (i.e., we will remove all art from the virtual galleries). In addition, we hypothesize that individuals primed to experience social connection prior to art exposure will experience lower perceived social disconnection and pain than those who are not primed.

DETAILED DESCRIPTION:
Research Design: 2 (virtual artwork exposure: present, absent) x 2 (prime: social connection prime: high, low) factorial experiment with a hanging control group (4 cells plus 1 control group, for a total of 5 cells) and 2 repeated measures. A priori power analysis using G*Power showed that the required sample size for a 5-group repeated measures experiment with 2 measurement times with 1-B error probability = .80 that expected small effect with a size of d = .10 and a significance level of p = .05 was a total of 305 participants (61 participants per cell).

Eligible individuals will be offered informed consent documentation via the StudyPages platform and then will be randomized to their study group:

1. Artwork present + Social connection prime high
2. Artwork present + Social connection prime low
3. Artwork absent + Social connection prime high
4. Artwork absent + Social connection prime low
5. Hanging control group - no exposure to any independent variables (i.e. artwork: present or absent; social connection prime: high or low)

Participants will fill out pre-intervention scales (pain intensity and unpleasantness; perceived social disconnection) prior to their virtual museum experience. Participants will then visit a virtual art museum gallery for 10 minutes or receive no exposure if they are in the hanging control group. In the artwork present condition, the virtual museum will feature paintings as part of an exhibition. In the artwork absent condition, paintings will be removed and thus the virtual museum will be empty. In the high social connection prime condition participants will be assigned to write an essay about a person and situation that made them feel valued, seen, and heard. In the low social connection prime condition participants will be assigned to write about a person and situation that made them feel ignored and not very valued. After 10 minutes within their condition participants will complete a post-intervention survey.

In addition, written responses to the social connection primes and museum visit data (e.g., user movement, object interaction, and perceptions about artwork in the museum) will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* read and write in English language
* chronic moderate to severe pain (≥ 6 months in duration; ≥ 4 in response to the question, "on average this week my pain intensity has been?" on a 0-10 NRS)
* lonely (≥ 4 on the 3-item Loneliness Scale)
* access to an electronic device with internet connection in order to participate in the study

Exclusion Criteria:

* dementia
* adults unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Social disconnection | Post-intervention (immediately)/Day 1
  Social disconnection scale; 12 items; scored 1 (not at all) - 5 (very much); range 12-60

SECONDARY OUTCOMES:
Pain unpleasantness | Post-intervention (immediately)/Day 1
  Numerical rating scale (NRS) score of 0 "not unpleasant" - 10 "Most unpleasant sensation imaginable ("intolerable")"
Pain intensity | Post-intervention (immediately)/Day 1
  Numerical rating scale (NRS) score of 0 "no pain" - 10 "worst pain imaginable"
Change in pain during intervention | Post-intervention (immediately)/Day 1
  Did you experience any pain relief during the museum experience? 1=Yes/0=No
Percent change in pain during intervention | Post-intervention (immediately)/Day 1
  If "Yes", what percent pain relief did you receive? 0%-100%
Perceptions of the artwork related to the positivity of the social world | Post-intervention (immediately)/Day 1
  The artwork in the museum made me feel (7-point likert scale anchored by "Negative about the social world" and "Positive about the social world")
Perceptions of the artwork related to connection to the social world | Post-intervention (immediately)/Day 1
  The artwork in the museum made me feel (7-point likert scale anchored by "Disconnected to the social world" and "Connected to the social world")
Perceptions of the artwork related to inclusion in the social world | Post-intervention (immediately)/Day 1
  The artwork in the museum made me feel (7-point likert scale anchored by "Excluded from the social world" and "Included in the social world")
Perceptions of the artwork related to positivity of social relationships | Post-intervention (immediately)/Day 1
  The artwork in the museum made me feel (7-point likert scale anchored by "Negative about my social relationships" and "Positive about my social relationships"

OTHER OUTCOMES:
Museum visit data - User Movement | During intervention
  Each user's avatar movement will be calculated in an x, y, z axis within the structure of the virtual museum.
Museum Visit Data - Object Interaction | During intervention
  Number of clicks on virtual museum artwork. Clicking gives users access to additional information about each piece of art.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No